CLINICAL TRIAL: NCT06037265
Title: First in Human Clinical Trial of the PAVmed PortIO Intraosseous Infusion System to Evaluate Safety and Performance
Brief Title: PR-0164 First in Human Clinical Trial of the PAVmed PortIO Intraosseous Infusion System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PAVmed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR-0164
Record Dates: First submitted 2023-08-29; First posted 2023-09-14 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Disease stage3; Chronic Kidney Disease stage4; Chronic Kidney Disease Stage 5; Poor Vascular Access
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Total Sample Size (Other): The total sample size will be up to 40 subjects that complete the full intended implant durations of either 7 days (n=up to 10) or60 days (n=up to 30). Group 1 patients will be enrolled first and at least 5 patients will complete the 7-day implant duration before Group 2 patients begin enrollment. Group 1 and Group 2 subjects can be screened in parallel. Group 2 enrollment will start immediately after at least 5 subjects in Group 1 have successfully completed the 7-day implantation period. Study subjects will have the PortIO device implanted by a qualified physician (Table 5) and then undergo prescribed, standard of care infusion regimen as determined by their treating physician over either the 7-day or the 60-day period. After the intended implant duration and use during the implant period, the device will then be removed and the subject will be followed for safety at 30 days after explant.
  Interventions: Device: PAVmed PortIO™ Intraosseous Infusion System

INTERVENTIONS:
Device: PAVmed PortIO™ Intraosseous Infusion System — The PortIO is intended to provide non-emergent vascular access in chronic kidney disease (CKD) patients where preservation of venous anatomy is desired and iatrogenic damage to the veins should be avoided and/or patients with poor/difficult vascular access. The PortIO device may be inserted into the proximal or distal tibia or the proximal humerus in adults, and provides up to 60 days of intraosseous vascular access for delivery of fluids and medications.

SUMMARY:
The PortIO is intended to provide non-emergent vascular access in chronic kidney disease (CKD) patients where preservation of venous anatomy is desired and iatrogenic damage to the veins should be avoided and/or patients with poor/difficult vascular access. The PortIO device may be inserted into the proximal or distal tibia or the proximal humerus in adults, and provides up to 60 days of intraosseous vascular access for delivery of fluids and medications.

DETAILED DESCRIPTION:
This is a prospective, open label, single arm, non-randomized, multicentric first in human clinical trial of the PortIO device for intraosseous infusion of fluids and/or medications for up to 60 days in subjects that meet the inclusion criteria. Both hospitalized patients as well as outpatients can be screened and, if appropriate, can be consented and enrolled into the study. They will have the PortIO device implanted by a qualified physician and then undergo prescribed infusions as needed and determined by the treating physician over either a 7-day or a 60-day period. The device will then be removed after the 7 days or 60 days of use and the subject followed up at 30 days after explant.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the following criteria are eligible for participation in the study:

  1. Subject is > 22 years old
  2. Subject has grade 3 or higher CKD and is receiving or may receive renal replacement therapy with hemodialysis OR has poor/difficult vascular access.
  3. Subject does NOT need urgent or emergent vascular access;
  4. Subject, or authorized representative, signs a written Informed Consent form to participate in the study, prior to any study mandated procedures
  5. Subject is willing and able to complete follow-up requirement

Exclusion Criteria:

* Subjects must be EXCLUDED from participation in this study if ANY of the following criteria are met:

  1. Fracture (within 6 months), bone tumor, or structural bone abnormality (such as osteogenesis imperfect, avascular necrosis, and severe osteoporosis) of the target bone
  2. Excessive overlying soft tissue, nerves, arteries, tendons or absence of anatomic landmarks at the target site
  3. Previous orthopedic procedure at or near the insertion site (e.g. artificial joint, rigid fixation hardware)
  4. IO access or attempted IO access in the target bone within 7 days
  5. Known or suspected allergy to any device component or materials contained in the device
  6. Local tissue factors preventing proper device stabilization and / or access including local infection, fragile tissue and absence of adequate or excessive overlying soft tissue.
  7. Subject with known unstable cardiac disease (recent MI within 30 days, cardiac surgery within 6 months, unstable angina, severe aortic stenosis/regurgitation, severe congestive heart failure, severe mitral stenosis/regurgitation), uncontrolled diabetes (blood glucose >240 mg/dl) or subjects on immunosuppressive medications (e.g. organ transplant patients)
  8. Subjects who are anticipated to receive infusion of blood or blood products, chemotherapeutic agents, hypertonic solutions, caustic agents or any agents known to harm bone marrow or cause bone marrow suppression such as azathioprine, procainamide, sulfasalazine via the test device.
  9. Insertion into the humerus on the same side as a previous mastectomy
  10. Known allergy to contrast media or local anesthetics (e.g. lidocaine, bupivacaine)
  11. Subjects with known bleeding disorders including thrombocytopenia, thrombasthenia, hemophilia or Von Willebrand's disease.
  12. Subjects with a history of hypercoagulable disorders such as protein S or C deficiency, Factor 5 Leiden resistance, Antithrombin III deficiency, Antiphospholipid antibody syndrome, Heparin Induced Thrombocytopenia etc.
  13. Subjects who are anticipated to need power injections via the test device for CT scan or angiography
  14. Subject has other medical, social or psychological problem that in the opinion of the investigator precludes them from fully participating
  15. Women who are pregnant, women who are attempting to become pregnant, as well as women who are breast feeding.

Ages: 22 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Primary Performance | Entire duration of Study an average of 2 years
  Incidence of successful implant in the target anatomic location; Patency through the implant duration, with final patency assessment performed immediately prior to device explant; Incidence of successful device explant
Primary Safety | Entire duration of Study and average of 2 years
  Incidence of serious device-related adverse events

SECONDARY OUTCOMES:
Secondary Endpoint | Entire duration of Study an average of 2 years
  Incidence of all device-related adverse events, whether serious or non-serious

CONTACTS AND LOCATIONS:
Overall Officials: Gisella Lopez, Study Director — Lucid Diagnostics
Locations (4):
- Colombia (4):
  - Cediul, Barranquilla, Atlántico
  - Sabbag Radiologos, Barranquilla, Atlántico
  - Cirulaser Andes, Bogotá, Bogota D.C.
  - Centro Medico Imbanaco, Cali, Valle de Cauca

IPD SHARING:
Plan to Share IPD: No